CLINICAL TRIAL: NCT07058740
Title: Safety and Feasibility of Early T-tube Cholangiography Performed Within 2 to 3 Days After LCBDE
Brief Title: Safety and Feasibility of Early T-tube Cholangiography Performed Within 2 to 3 Days After Laparoscopic Common Bile Duct Exploration
Acronym: LCBDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Piyou Ji (Other)
Responsible Party: Sponsor-Investigator, Piyou Ji, associate chief physician, Yantai Affiliated Hospital of Binzhou Medical University
Organization: Yantai Affiliated Hospital of Binzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F-KY-0022-20220325-01
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Common Bile Duct Calculi; Laparoscopic Abdominal Surgery; Cholangiography
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early cholangiography group (Experimental): T-tube cholangiography performed 2-3 days postoperatively
  Interventions: Procedure: early cholangiography
- delayed cholangiography group (No Intervention): T-tube cholangiography performed >3 days postoperatively

INTERVENTIONS:
Procedure: early cholangiography — We perform cholangiography on the early group in advance
  Arms: early cholangiography group

SUMMARY:
Current clinical evidence indicates that 10-20% of patients with symptomatic cholelithiasis present with concomitant common bile duct stones (CBDS), a clinical scenario requiring tailored therapeutic approaches. In contemporary surgical practice, laparoscopic common bile duct exploration (LCBDE) combined with T-tube drainage (TTD) has emerged as the intervention of choice for complex biliary pathologies. This approach demonstrates particular efficacy in managing three distinct clinical categories: acute infective conditions such as suppurative cholangitis, structural anomalies including biliary tract injuries and sphincter of Oddi dysfunction, and post-interventional complications spanning biliary strictures, unsuccessful endoscopic retrograde cholangiopancreatography (ERCP) attempts, and significant inflammatory changes in the ductal architecture.

The T-tube serves multiple functions with significant clinical implications. Its primary roles include: (1) enabling intra- and postoperative cholangiography to detect residual stones or clarify biliary anatomy; (2) facilitating bile drainage to reduce ductal pressure and postoperative bile leakage risks; (3) providing a "window" for monitoring biliary secretion, which helps in assessing biliary function and recovery; (4) establishing a sinus tract for secondary stone retrieval, thereby enhancing therapeutic efficacy. T-tubes play a vital role in biliary disease management due to their proven safety and functional advantages in post-LCBDE care.

Postoperative T-tube cholangiography was routinely obtained prior to biliary drainage occlusion to definitively exclude residual choledocholithiasis and confirm contrast agent passage into the duodenum in patients undergoing LCBDE with TTD. While T-tube cholangiography provides crucial postoperative evaluation, it may also lead to complications such as abdominal pain, fever, diarrhea, and bile leakage around the T-tube. The smooth flow of contrast agent into the duodenum during cholangiography is a key criterion for determining whether the T-tube can be clamped. Once this condition is met, the T-tube can be closed, and the drainage bag removed, minimizing the impact on daily activities and marking a significant phase in postoperative recovery.

The timing of T-tube cholangiography directly affects the duration of drainage bag use, but there is no consensus on the earliest timing in clinical practice. Most studies recommend performing cholangiography at least 5 days postoperatively. Zhang et al. reported performing cholangiography 5 days postoperatively, while four other studies consistently chose 7 days postoperatively. Additionally, K. S. Gurusamy suggest performing cholangiography 10 to 14 days postoperatively. The earliest timing for postoperative T-tube cholangiography remains unclear and requires further research to guide clinical practice.

To evaluate the safety and feasibility of early post-LCBDE T-tube cholangiography (2-3days), this retrospective cohort study compared patients receiving biliary imaging within the early window (≤3days) versus those undergoing delayed protocol (>3days postoperatively).Furthermore, the data from patients who underwent cholangiography within 2-3 days were compared with data from other studies to assess the clinical outcomes and potential complications of early T-tube cholangiography, aiming to optimize postoperative management strategies.

ELIGIBILITY:
Inclusion Criteria:

* 1.Confirmed diagnosis of CBDS; 2.LCBDE with T-tube placement; 3.Postoperative T-tube cholangiography.

Exclusion Criteria:

* 1.Incomplete data; 2.Animal or non-human studies; 3.Case reports or single-case studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
hospital stay | From enrollment to the end of treatment at 2 weeks
  patients stay in hospital after operations
complications | From enrollment to the end of treatment at 4 weeks
  bile leak and pancreatitis

CONTACTS AND LOCATIONS:
Locations (1):
- Yantai affiliated hospital of Binzhou Medical University, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes